CLINICAL TRIAL: NCT03246074
Title: Phase I Clinical Trial of Combined Fostamatinib and Paclitaxel in Ovarian Cancer
Brief Title: Clinical Trial of Combined Fostamatinib and Paclitaxel in Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Rigel Pharmaceuticals (Industry); Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1708; IRB00271541 (Other: JHM IRB)
Record Dates: First submitted 2017-06-15; First posted 2017-08-11 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer
Keywords: Phase I; Ovarian Cancer; Fostamatinib and Paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fostamatinib; BID protein, human; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fostamatinib 100 mg bid and Paclitaxel (Experimental): Participants will receive paclitaxel on Days 1, 8 and 15 of each cycle and fostamatinib at a fixed oral dose of 100mg twice daily throughout each 28-day cycle.
  Interventions: Drug: Fostamatinib 100 mg bid and Paclitaxel
- Fostamatinib 150 mg bid and Paclitaxel (Experimental): Participants will receive paclitaxel on Days 1, 8 and 15 of each cycle and fostamatinib at a fixed oral dose of 150mg twice daily throughout each 28-day cycle.
  Interventions: Drug: Fostamatinib 150 mg bid and Paclitaxel
- Fostamatinib 200 mg bid and Paclitaxel (Experimental): Participants will receive paclitaxel on Days 1, 8 and 15 of each cycle and fostamatinib at a fixed oral dose of 150mg twice daily throughout each 28-day cycle.
  Interventions: Drug: Fostamatinib 200 mg bid and Paclitaxel

INTERVENTIONS:
Drug: Fostamatinib 100 mg bid and Paclitaxel — Drug: Fostamatinib (oral; 100 mg bid)
  Drug: Paclitaxel (60-80 mg/m2)
  Other Names: Fostamatinib and Abraxane
  Arms: Fostamatinib 100 mg bid and Paclitaxel
Drug: Fostamatinib 150 mg bid and Paclitaxel — Drug: Fostamatinib (oral; 150 mg bid)
  Drug: Paclitaxel (60-80 mg/m2)
  Other Names: Fostamatinib and Abraxane
  Arms: Fostamatinib 150 mg bid and Paclitaxel
Drug: Fostamatinib 200 mg bid and Paclitaxel — Drug: Fostamatinib (oral; 200 mg bid)
  Drug: Paclitaxel (60-80 mg/m2)
  Other Names: Fostamatinib and Abraxane
  Arms: Fostamatinib 200 mg bid and Paclitaxel

SUMMARY:
This research is being done to test the safety of the combination of the study drugs fostamatinib and paclitaxel. This study tests different doses of the drugs to see which doses are safest in people with ovarian cancer when given together.

DETAILED DESCRIPTION:
This is a phase I, open-label, non-randomized multicenter dose-escalation study with the primary objective to determine the maximally tolerated dose (MTD) of fostamatinib when administered with weekly paclitaxel in women with recurrent platinum-resistant ovarian, fallopian tube, or primary peritoneal cancer.

Between 8 and 18 adult female subjects will be enrolled and receive weekly paclitaxel in combination with increasing doses of fostamatinib. There will be three dosing regimens of fostamatinib (100 mg bid, 150 mg bid, and 200mg bid) selected based on the FDA approved doses and prior phase I studies of single agent fostamatinib. Dose-escalation will follow a modified toxicity probability interval (mTPI) design. In this study, up to 18 adult female subjects will be enrolled and receive weekly paclitaxel in combination with fostamatinib at the MTD of the combination; at least 6 patients will receive fostamatinib plus paclitaxel at the MTD. A total of up to 30 patients will be enrolled in this study.

ELIGIBILITY:
* Inclusion Criteria

  1. Patients must have histologically or cytologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. Histologic documentation (via the pathology report) of the original primary tumor is required.
  2. Patients must have measurable disease, according to RECIST v1.1.
  3. Patients must have recurrent, platinum-resistant disease (defined as having relapsed within 6 months of last platinum-containing regimen) or be unable to receive further platinum therapy. There is no limit on the number of prior treatment regimens; however, patients may not have previously received weekly paclitaxel in the recurrent setting. Previous dose dense paclitaxel as initial therapy is allowable.
  4. Patients must have the ability to take oral medications.
  5. Females, age ≥18 years.
  6. ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
  7. Life expectancy of greater than 3 months.
  8. Patients must have normal organ and marrow function.
  9. Patients with a diagnosis of hypertension are required to have adequate blood pressure control prior to enrollment, defined as blood pressure ≤ 140/90 mmHg.
  10. The effects of fostamatinib on the developing human fetus are unknown. For this reason, women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
  11. Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial if the anti-retroviral therapy is not an excluded concurrent medication.
  12. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated and the suppressive therapy is not an excluded concurrent medication.
  13. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load and the HCV therapy is not an excluded concurrent medication.
  14. Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
  15. Patients who are willing and able to comply with the protocol and study procedures.

      Tumor biopsy or paracentesis for tumor cells before therapy (at baseline) and after initiation of treatment (before Cycle 2) for at least 75% of subjects if this is clinically and safely feasible to do so. For patients who have had tumor tissue sampled within 6 months of enrollment and no intervening anti-neoplastic therapy, archived tissue may satisfy the requirement of the pre-treatment biopsy with permission of the protocol chair.
  16. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial, with permission of the protocol chair.
  17. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
  18. The effects of fostamatinib on the developing human fetus are unknown. For this reason and because spleen tyrosine kinase inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  19. Ability to understand and the willingness to sign a written informed consent document.
* Exclusion Criteria

  1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study. Hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration.
  2. Patients who have not recovered (CTCAE v4.03 grade ≤1) from adverse events due to agents administered more than 4 weeks earlier, unless those events are deemed to have returned to baseline, are irreversible, or are unlikely to develop into a life-threatening condition at the permission of the Protocol Chair (e.g., alopecia).
  3. Patients who are currently receiving or have previously received any other investigational agents within 3 weeks prior to entering the study.
  4. Patients with known untreated brain metastases, as progressive neurologic dysfunction may develop that would confound the evaluation of neurologic and other adverse events.
  5. Patients with Grade 2 or greater neuropathy.
  6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to fostamatinib or paclitaxel. Patients who are able to tolerate paclitaxel on a desensitization protocol will be allowed.
  7. Strong CYP3A4 inhibitors or inducers should not be used within 3 days of Day 1 dosing until the end of study. Moderate CYP3A4 inhibitors or inducers should be used with caution.
  8. Uncontrolled intercurrent illness
  9. Pregnant women are excluded from this study because the potential for teratogenic or abortifacient effects of fostamatinib are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with fostamatinib, breastfeeding should be discontinued if the mother is treated with fostamatinib. These potential risks may also apply to other agents used in this study.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must have ovarian, fallopian tube or peritoneal carcinoma.
Enrollment: 35 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Gaillard, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 participants were consented. 8 were screen failures. 27 were assigned to study arms.
Groups:
- Fostamatinib 100 mg Bid and Paclitaxel: Participants will receive paclitaxel on Days 1, 8 and 15 of each cycle and fostamatinib at a fixed oral dose of 100mg twice daily throughout each 28-day cycle.
  Fostamatinib 100 mg bid and Paclitaxel: Drug: Fostamatinib (oral; 100 mg bid)
  Drug: Paclitaxel (60-80 mg/m2)
- Fostamatinib 150 mg Bid and Paclitaxel: Participants will receive paclitaxel on Days 1, 8 and 15 of each cycle and fostamatinib at a fixed oral dose of 150mg twice daily throughout each 28-day cycle.
  Fostamatinib 150 mg bid and Paclitaxel: Drug: Fostamatinib (oral; 150 mg bid)
  Drug: Paclitaxel (60-80 mg/m2)
- Fostamatinib 200 mg Bid and Paclitaxel: Participants will receive paclitaxel on Days 1, 8 and 15 of each cycle and fostamatinib at a fixed oral dose of 150mg twice daily throughout each 28-day cycle.
  Fostamatinib 200 mg bid and Paclitaxel: Drug: Fostamatinib (oral; 200 mg bid)
  Drug: Paclitaxel (60-80 mg/m2)
Period: Overall Study
Arm/Group | Fostamatinib 100 mg Bid and Paclitaxel | Fostamatinib 150 mg Bid and Paclitaxel | Fostamatinib 200 mg Bid and Paclitaxel
Started | 6 | 3 | 18
Completed | 6 | 3 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostamatinib 100 mg Bid and Paclitaxel | Fostamatinib 150 mg Bid and Paclitaxel | Fostamatinib 200 mg Bid and Paclitaxel | Total
Number analyzed (Participants) | 6 | 3 | 18 | 27
Age, Continuous [Median (Full Range); unit: years] | 62.9 [40.9 to 75.4] | 62.1 [37.9 to 72.4] | 62.0 [35.5 to 79.7] | 62.12 [35.47 to 79.73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 18 | 27
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 5 | 3 | 17 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 5 | 5
  White | 5 | 2 | 10 | 17
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Fostamatinib
Description: The number of dose limiting toxicities (DLTs) at each dose level will be reported. All toxicities will be reported by type and grade using NCI CTCAE version 4.03.
Time Frame: First cycle (28 days) of treatment
Measure: Number; unit: Dose Limiting Toxicities (DLTs)
Arm/Group | Fostamatinib 100 mg Bid and Paclitaxel | Fostamatinib 150 mg Bid and Paclitaxel | Fostamatinib 200 mg Bid and Paclitaxel
Number analyzed (Participants) | 6 | 3 | 18
Dose Limiting Toxicities (DLTs) | 0 | 0 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Fostamatinib
Description: The MTD will be determined as the dose level with the highest probability of having a risk of DLT in the acceptable region based on the mTPI dose-escalation design. Measured at 28 days (DLT period).
Time Frame: 28 days
Population: Participants included in the dose-escalation are reported
Measure: Number; unit: milligrams
Groups:
- Participants in Dose-escalation Portion of the Trial, Either at the 100, 150 or 200mg Bid Dose Level: The primary objective was determine the maximally tolerated dose (MTD) of fostamatinib when administered with weekly paclitaxel. The design included three dose levels of fostamatinib, 100, 150, and 200 mg of fostamatinib with a fixed dosage of paclitaxel at each. Dose escalation followed a modified toxicity probability interval (mTPI) design.
Arm/Group | Participants in Dose-escalation Portion of the Trial, Either at the 100, 150 or 200mg Bid Dose Level
Number analyzed (Participants) | 12
milligrams | 200

3. Secondary Outcome: Objective Response Rate in the Study Population Treated With the Combination of Fostamatinib and Paclitaxel
Description: Number of participants within each objective response as seen on imaging/RECIST 1.1. Per response evaluation criteria in solid tumors criteria (RECIST v1.1) for target lesions: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- All Participants Treated With Fostamatinib and Paclitaxel at 100mg BID; All Participants Treated With Fostamatinib and Paclitaxel at 150mg BID; All Participants Treated With Fostamatinib and Paclitaxel at 200mg BID: Only those subjects who have measurable disease present at baseline, have received at least 1 cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response.
Arm/Group | All Participants Treated With Fostamatinib and Paclitaxel at 100mg BID | All Participants Treated With Fostamatinib and Paclitaxel at 150mg BID | All Participants Treated With Fostamatinib and Paclitaxel at 200mg BID
Number analyzed (Participants) | 6 | 3 | 18
Participants
  Partial Response (PR) | 1 | 0 | 7
  Stable Disease (SD) | 0 | 1 | 5
  Progressive Disease (PD) | 1 | 2 | 4
  Non-Evaluable (NE) | 4 | 0 | 2

4. Secondary Outcome: Progression-free Survival in the Study Population Treated With the Combination of Fostamatinib and Paclitaxel
Description: Progression-free survival (PFS) will be described by the method of Kaplan and Meier. Median PFS in months will be estimated along with its 95% confidence interval. Per response evaluation criteria in solid tumors (RECIST v1.1), Progressive Disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants Treated With Fostamatinib and Paclitaxel at 100mg BID | All Participants Treated With Fostamatinib and Paclitaxel at 150mg BID | All Participants Treated With Fostamatinib and Paclitaxel at 200mg BID
Number analyzed (Participants) | 6 | 3 | 18
Months | 1.445 [0.92 to NA] — Value is reported as NA because its estimate (from Greenwood's Formula and asymptotic normal distribution assumption) is larger than 1 (outside the range between 0 and 1). | 1.81 [1.22 to NA] — Value is reported as NA because its estimate (from Greenwood's Formula and asymptotic normal distribution assumption) is larger than 1 (outside the range between 0 and 1). | 4.305 [2.69 to 6.37]

5. Secondary Outcome: Pharmacokinetic (PK) Profile of Fostamatinib When Combined With Weekly Paclitaxel - Tmax
Description: Tmax (hours) was used to summarize pharmacokinetic marker profile for fostamatinib. Tmax (hours): Time to reach maximum plasma concentration of R406, the active meta
Time Frame: First cycle (28 days) of treatment
Population: 1 patient at the 100 mg dose and 1 patient at the 200 mg did not have all PKs drawn and were not included in the PK analysis
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fostamatinib 100 mg Bid and Paclitaxel | Fostamatinib 150 mg Bid and Paclitaxel | Fostamatinib 200 mg Bid and Paclitaxel
Number analyzed (Participants) | 5 | 3 | 17
hours | 1.96 (2.26) | 1.69 (1.13) | 1.9 (1.10)

6. Secondary Outcome: Pharmacokinetic (PK) Profile of Fostamatinib When Combined With Weekly Paclitaxel - Cmax
Description: Cmax (ng/mL) was used to summarize pharmacokinetic marker profile for fostamatinib. Cmax (ng/mL): Maximum plasma concentration of R406.
Time Frame: First cycle (28 days) of treatment
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/ML
Arm/Group | Fostamatinib 100 mg Bid and Paclitaxel | Fostamatinib 150 mg Bid and Paclitaxel | Fostamatinib 200 mg Bid and Paclitaxel
Number analyzed (Participants) | 5 | 3 | 17
ng/ML | 803.4 (452.0) | 1309.3 (599.7) | 1187.2 (784.0)

7. Secondary Outcome: Pharmacokinetic (PK) Profile of Fostamatinib When Combined With Weekly Paclitaxel - Area Under the Curve (AUC) 0-6hours
Description: AUC0-6h (ng*h/mL) was used to summarize pharmacokinetic marker profile for fostamatinib. AUC0-6h (ng*h/mL): Area under the concentration-time curve for R406 up to 6 hours post-dosing.
Time Frame: First cycle (28 days) of treatment
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Fostamatinib 100 mg Bid and Paclitaxel | Fostamatinib 150 mg Bid and Paclitaxel | Fostamatinib 200 mg Bid and Paclitaxel
Number analyzed (Participants) | 5 | 3 | 17
ng*h/mL | 2265.7 (1328.7) | 4067.3 (1177.8) | 3958.8 (2104.1)

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of first dose of study drug to 30 days after the last dose, up to 55 weeks.
Arm/Group | Fostamatinib 100 mg Bid and Paclitaxel | Fostamatinib 150 mg Bid and Paclitaxel | Fostamatinib 200 mg Bid and Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 1/18
Serious Adverse Events (participants affected / at risk) | 3/6 | 0/3 | 7/18
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fostamatinib 100 mg Bid and Paclitaxel (N=6) | Fostamatinib 150 mg Bid and Paclitaxel (N=3) | Fostamatinib 200 mg Bid and Paclitaxel (N=18)
Abdominal infection (Infections and infestations) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fostamatinib 100 mg Bid and Paclitaxel (N=6) | Fostamatinib 150 mg Bid and Paclitaxel (N=3) | Fostamatinib 200 mg Bid and Paclitaxel (N=18)
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 2 | 14
Nausea (Gastrointestinal disorders) | 3 | 2 | 10
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 7
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 6
Vomiting (Gastrointestinal disorders) | 2 | 0 | 4
Constipation (Gastrointestinal disorders) | 0 | 0 | 4
Bloating (Gastrointestinal disorders) | 1 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1
Edema limbs (General disorders) | 0 | 2 | 3
Fatigue (General disorders) | 2 | 2 | 11
Fever (General disorders) | 1 | 0 | 7
Non-cardiac chest pain (General disorders) | 2 | 0 | 3
Pain (General disorders) | 2 | 1 | 4
Localized edema (General disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 9
Dysgeusia (Nervous system disorders) | 1 | 1 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 5
Presyncope (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 3
Ataxia (Nervous system disorders) | 0 | 0 | 1
Concentration impairment (Nervous system disorders) | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 9
Alanine aminotransferase increased (Investigations) | 2 | 0 | 4
Weight gain (Investigations) | 0 | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 3
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Creatinine increased (Investigations) | 1 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 3
Weight loss (Investigations) | 0 | 0 | 2
Urine output decreased (Investigations) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 5
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 4
Abdominal infection (Infections and infestations) | 1 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 0 | 2
Skin infection (Infections and infestations) | 0 | 0 | 2
Bronchial infection (Infections and infestations) | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hpercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 6
Thromboembolic event (Vascular disorders) | 1 | 0 | 3
Chest pain- cardiac (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT03246074/Prot_SAP_000.pdf